CLINICAL TRIAL: NCT00990301
Title: A Study to Compare the Relative Bioavailability of Moexipril HCl/Hydrochlorothiazide 15mg/25mg Tablets (Paddock Laboratories, Inc) and Uniretic® 15mg/25mg Tablets (Schwarz Pharma)(Moexipril HCl/Hydrochlorothiazide) in Healthy Adult Volunteers Under Fasting Conditions.
Brief Title: A Study to Compare the Relative Bioavailability of Moexipril HCl/Hydrochlorothiazide in Healthy Adult Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Paddock Laboratories, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10630201
Record Dates: First submitted 2009-10-04; First posted 2009-10-06 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Healthy
Keywords: Healthy Subjects; Bioequivalence
MeSH Terms: interventions — moexipril; Hydrochlorothiazide; Tablets

ARMS (2):
- Moexipril HCl/ Hydrochlorothiazide 15mg/25mg Tablets (Experimental)
  Interventions: Drug: Moexipril HCl/ Hydrochlorothiazide 15mg/ 25mg Tablet, Paddock Laboratories, Inc.
- Uniretic® 15mg/25mg Tablets (Active Comparator)
  Interventions: Drug: Moexipril HCl/ Hydrochlorothiazide 15mg/ 25mg Tablet, Paddock Laboratories, Inc.; Drug: Uniretic® 15mg/25mg Tablets

INTERVENTIONS:
Drug: Moexipril HCl/ Hydrochlorothiazide 15mg/ 25mg Tablet, Paddock Laboratories, Inc. — test drug
Drug: Uniretic® 15mg/25mg Tablets — reference drug
  Arms: Uniretic® 15mg/25mg Tablets

SUMMARY:
The purpose of this study was to evaluate the relative bioavailability of Paddock Laboratories, Inc.'s test formulation of Moexipril/ Hydrochlorothiazide 15mg/25mg tablets with a reference formulation Uniretic®(Moexipril/ Hydrochlorothiazide) 15mg/25mg tablets, under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening

Exclusion Criteria:

* Positive test results for HIV or Hepatitis B or C
* History of allergy or sensitivity to Moexipril, Hydrochlorothiazide or related drugs

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)

PRIMARY OUTCOMES:
Bioequivalence specified outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Kennedy, M.D., Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Pittsburgh, Pennsylvania, United States